CLINICAL TRIAL: NCT05992155
Title: An Open-Label, Phase 1 Study to Compare Pharmacokinetics, Safety, and Tolerability of a Single Oral Dose of TAK-279 in Subjects With or Without Renal Impairment
Brief Title: A Study of TAK-279 in Adults With or Without Kidney Problems
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TAK-279-1003
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Renal Impairment; Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1, Severe RI: TAK-279 50 mg (Experimental): Participants with severe RI will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part A of the study.
  Interventions: Drug: TAK-279
- Cohort 2, Normal Renal Function: TAK-279 50 mg (Experimental): Participants with normal renal function will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part A of the study.
  Interventions: Drug: TAK-279
- Cohort 3, Moderate RI: TAK-279 50 mg (Experimental): Participants with moderate RI will receive a single oral dose of TAK-279 50 mg, on Day 1 in Part B of the study.
  Interventions: Drug: TAK-279

INTERVENTIONS:
Drug: TAK-279 — TAK-279 capsules.

SUMMARY:
The main aim of this study is to find out how the body processes 1 dose of TAK-279 (pharmacokinetics) in participants with kidney problems compared to participants without kidney problems. Other aims are to check for side effects from TAK-279 and to learn how well participants tolerate 1 dose of TAK-279.

The participants will need to stay at the clinic for 11 days.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-279. TAK-279 is being tested to assess the pharmacokinetics (PK), safety, and tolerability of TAK-279 in participants with severe (Part A) and moderate (Part B) renal impairment (RI) compared to healthy participants with normal renal function.

The study will enroll up to 48 patients. Participants will be assigned to following study cohorts in Parts A and B to receive single-dose of TAK-279:

* Cohort 1, Severe RI (12 participants): TAK-279 50 mg
* Cohort 2, Normal Renal Function (12 to 24 participants): TAK-279 50 mg
* Cohort 3, Moderate RI (12 participants): TAK-279 50 mg

If the decision to proceed to Part B is made, participants with moderate RI will be enrolled in Cohort 3 of the study. Participants in Cohort 3 will receive single-dose of TAK-279 50 mg and will be compared with the participants who meet the matching criteria of Cohort 2 with normal renal function. A participant with normal renal function (either from Part A or enrolled in Part B) may be matched to only one participant with RI in Part B.

This multi-center trial will be conducted in the United States. The overall duration of the study is up to 44 days. Participants will be followed up for 14 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

A. Participants with RI:

The participants must fulfill the following inclusion criteria to be eligible for participation in the study (participants who do not qualify based on a reversible condition or mild intercurrent illness may be re-screened after the condition is resolved. Screening tests may be repeated if in the Investigator's opinion the test needs to be repeated):

1. Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.
2. Adult male or female participant aged ≥18 years, at screening.
3. Has a body weight greater than 50 kg and has a body mass index (BMI) ≥18.0 and ≤39.0 kilograms per meters squared (kg/m^2), at screening.
4. Continuous non-smoker or moderate smoker (≤10 cigarettes/day or the equivalent [including electronic cigarettes]) before screening. Participant must agree to smoke no more than 5 cigarettes or equivalent/day (including electronic cigarettes) from the 7 days prior to TAK-279 dosing.
5. Aside from RI, be sufficiently healthy for study participation based upon medical history, physical examination, vital signs, electrocardiograms (ECGs), and screening clinical laboratory profiles, as deemed by the Investigator or designee, including:

   * Supine blood pressure (BP) is ≥90/40 mmHg (asymptomatic) and ≤180/100 mmHg, at screening;
   * Supine pulse rate (PR) is ≥40 beats per minute (bpm) and ≤99 bpm, at screening;
   * Liver function tests including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin within the upper limit of normal (ULN) at screening and at check-in.
   * Creatine phosphokinase (CPK) ≤ ULN at the screening visit and at check-in.
   * Amylase and lipase ≤ ULN at the screening visit and at check-in.
6. Estimated glomerular filtration rate (eGFR) based on the Modification of Diet in Renal Disease (MDRD) equation at screening as follows,

   * Severe RI: <30 milliliters per minute (mL/min), not on dialysis;
   * Moderate RI: 30-59 mL/min.
7. Has chronic RI for at least 3 months before screening, and the RI must be stable, i.e., no significant changes (i.e., ≥30%) in renal function in the 30 days preceding screening (or since the last visit if within 6 months before screening) and treatment with stable doses of medication.
8. Female participants of childbearing potential agree to comply with highly effective contraceptive requirements of the protocol.
9. Male participants must agree to comply with effective contraceptive requirements of the protocol.

B. Healthy Participants:

1. Understands the study procedures in the ICF, and be willing and able to comply with the protocol.
2. Adult male or female participants aged ≥18 years, at screening. Participant will be matched by age (±10 years) and sex to a participant with severe RI (Part A) and/or a participant with moderate RI (Part B).
3. Has a body weight greater than 50 kg and has a BMI ≥18.0 and ≤39.0 kg/m2, at screening. Participant will be matched by body weight (±15 kg) to a participant with severe RI (Part A) and/or a participant with moderate RI (Part B).
4. Continuous non-smoker or moderate smoker (≤10 cigarettes/day or the equivalent [including electronic cigarettes]) before screening. Participant must agree to smoke no more than 5 cigarettes or equivalent/day (including electronic cigarettes) from the 7 days prior to TAK-279 dosing.
5. Medically healthy with no clinically significant medical history, physical examination, vital signs, ECGs, and screening clinical laboratory profiles, as deemed by the Investigator or designee, including:

   * Supine BP is ≥90/40 mmHg and ≤150/95 mmHg, at screening;
   * Supine PR is ≥40 bpm and ≤99 bpm, at screening;
   * Liver function tests including ALT, AST, ALP, and total bilirubin within ULN at screening and at check-in.
   * CPK ≤ ULN at the screening visit and at check-in.
   * Amylase and lipase ≤ ULN at the screening visit and at check-in.
6. eGFR based on the MDRD equation at screening as follows:

   * Normal renal function: ≥90 mL/min.
7. Female participants of childbearing potential agree to comply with highly effective contraceptive requirements of the protocol.
8. Male participants must agree to comply with effective contraceptive requirements of the protocol.

Exclusion Criteria:

A. Participants with RI:

The participant must be excluded from participating in the study if the participant:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of screening or expected during the conduct of the study.
2. Has history or presence of clinically significant medical or psychiatric condition or disease (aside from RI) in the opinion of the Investigator or designee.
3. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to dosing, as assessed by the Investigator or designee;
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to dosing;
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis);
   * An infected joint prosthesis unless that prosthesis has been removed or replaced within 60 days prior to dosing;
   * Opportunistic infections (eg, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis);
   * Cancer or lymphoproliferative disease with the exception of successfully treated nonmelanoma skin cancer (NMSC) or basal cell carcinoma and/or localized carcinoma in situ of the cervix;
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy;
5. Has had a failed renal transplant or a nephrectomy.
6. Has history or presence of alcoholism and/or drug abuse within the past 6 months prior to dosing, as determined by the Investigator or designee.
7. Has history or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
8. Female with a positive pregnancy test at screening or check-in or who is lactating.
9. Has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the study, in the opinion of the Investigator or designee.
10. Has positive results for the urine or saliva drug screen at screening or check-in, unless the positive drug screen is due to prescription drug use that is approved by the Investigator or designee and Sponsor.
11. Has positive results for urine or breath alcohol screen at screening or check-in.
12. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) for the prohibited time period.
13. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
14. Has made a donation of blood or had significant blood loss within 56 days prior to dosing.
15. Has made a plasma donation within 7 days prior to dosing.
16. Participated in another clinical study within 30 days prior to dosing. The 30-day window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
17. Herpes infections:

    * Has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day -1.
    * History of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
18. Positive results for non-herpetic viral diseases at screening:

    * Hepatitis C virus (HCV) antibody and a positive confirmatory test result for HCV ribonucleic acid (RNA) (nucleic acid test or polymerase chain reaction (PCR));
    * Hepatitis B surface antigen (HBsAg)+, hepatitis B virus deoxyribonucleic acid (DNA), or anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody (HBcAb+ and HBsAb-);
    * Human immunodeficiency virus (HIV).
19. Tuberculosis (TB):

    * History of active TB infection, regardless of treatment status;
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the Investigator or designee;
    * Has evidence of latent tuberculosis infection (LTBI) as evidenced by a positive QuantiFERON-TB Gold (QFT) result OR 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis; Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines);
    * Has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.

B. For Healthy Participants:

The participant must be excluded from participating in the study if the participant:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of screening or expected during the conduct of the study.
2. Has history or presence of clinically significant medical or psychiatric condition or disease in the opinion of the Investigator or designee.
3. Has history of any illness that, in the opinion of the Investigator or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
4. Has a history of any of the following:

   * Active infection or febrile illness within 7 days prior to dosing, as assessed by the Investigator or designee.
   * Symptoms suggestive of systemic or invasive infection requiring hospitalization or treatment within 8 weeks prior to dosing.
   * Chronic or recurrent bacterial disease, including but not limited to chronic pyelonephritis or cystitis, chronic bronchitis/pneumonitis, osteomyelitis, or chronic skin ulcerations/infections or fungal infections (except superficial nailbed mycosis).
   * An infected joint prosthesis unless that prosthesis has been removed or replaced within 60 days prior to dosing.
   * Opportunistic infections (eg, Pneumocystis jirovecii pneumonia, histoplasmosis, coccidiomycosis).
   * Cancer or lymphoproliferative disease, with the exception of successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix.
   * Known or suspected condition/illness that is consistent with compromised immunity, including but not limited to any identified congenital or acquired immunodeficiency; splenectomy.
5. Has history or presence of alcoholism and/or drug abuse within the past 2 years prior to dosing, as determined by the Investigator or designee.
6. Has history or presence of clinically significant hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
7. Female with a positive pregnancy test at screening or check-in, or who is lactating.
8. Has ECG abnormalities that are considered clinically significant and would pose an unacceptable risk to the participant if he or she participated in the study, in the opinion of the Investigator or designee.
9. Has positive results for the urine or saliva drug screen at screening or check-in, unless the positive drug screen is due to prescription drug use that is approved by the Investigator or designee and Sponsor.
10. Has positive results for urine or breath alcohol screen at screening or check-in.
11. Unable to refrain from or anticipates the use of any medication or substance (including prescription or over-the-counter, vitamin supplements, natural or herbal supplements) for the prohibited time period.
12. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to dosing and throughout the study.
13. Has made a donation of blood or had significant blood loss within 56 days prior to dosing.
14. Has made a plasma donation within 7 days prior to dosing.
15. Participated in another clinical study within 30 days prior to dosing. The 30-day window will be derived from the date of the last dosing in the previous study to Day 1 of the current study.
16. Herpes infections:

    * Has active herpes virus infection, including herpes zoster or herpes simplex 1 and 2 (demonstrated on physical examination and/or medical history) at screening or Day -1.
    * History of serious herpetic infection that includes any episode of disseminated disease, multidermatomal herpes zoster virus, herpes encephalitis, ophthalmic herpes, or recurrent herpes zoster (defined as 2 episodes within 2 years).
17. Positive results for non-herpetic viral diseases at screening:

    * HCV antibody and a positive confirmatory test result for HCV RNA (nucleic acid test or PCR);
    * HBsAg+, hepatitis B virus DNA, or anti-hepatitis B core antibody without concurrent positive hepatitis B surface antibody (HBcAb+ and HBsAb-);
    * HIV.
18. TB:

    * History of active TB infection, regardless of treatment status;
    * Has signs or symptoms of active TB (including but not limited to chronic fever, chronic productive cough, night sweats, or weight loss) as judged by the Investigator or designee;
    * Has evidence of LTBI as evidenced by a positive QFT result OR 2 indeterminant QFT results and does not have documentation of appropriate LTBI prophylaxis. Participant remains eligible if he or she can provide documentation of prior and complete treatment for LTBI (appropriate in duration and type per current local country guidelines);
    * Has had any imaging study during or 6 months prior to screening, including x-ray, chest computed tomography, magnetic resonance imaging, or other chest imaging suggesting evidence of current active or a history of active TB.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum Observed Plasma Concentration for TAK-279 | Predose to Day 10
AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-279 | Predose to Day 10
AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for TAK-279 | Predose to Day 10

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | From study start through 14 days after last dose administration (up to approximately 42 days)
  An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Number of Participants With Adverse Events of Special Interest (AESIs) | From study start through 14 days after last dose administration (up to approximately 42 days)
Number of Participants With Markedly Abnormal Values for Vital Signs | Up to Day 10
Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings | Up to Day 10
Number of Participants With Markedly Abnormal Laboratory Values | Up to Day 10
Number of Participants With Clinically Significant Physical Examination Findings | Up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Research by Design, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link — https://clinicaltrials.takeda.com/study-detail/384ecc6960fc4129?idFilter=%5B%22TAK-279-1003%22%5D